CLINICAL TRIAL: NCT03816761
Title: An Exploratory Trial Investigating the Safety and Efficacy of Fast-acting Insulin Aspart in a Closed-loop Insulin Delivery System (Bionic Pancreas) in Adults With Type 1 Diabetes
Brief Title: Research Study to Look at Fast-acting Insulin Aspart With the Insulin Pump System 'iLet™' in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-4360; U1111-1205-1788 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Fast-acting insulin aspart, default tmax setting (Experimental): Participants will receive fast-acting insulin aspart using the iLet™ with default tmax setting (t65 = 65 minutes) in two different treatment periods in a cross-over manner. There will be 3 different cohorts with 2 treatment periods in each cohort.
  Interventions: Drug: Fast-acting insulin aspart; Device: iLet™
- Fast-acting insulin aspart, non-default tmax setting (Experimental): Participants will receive fast-acting insulin aspart using the iLet™ with non-default tmax setting (t50 = 50 minutes, t40 = 40 minutes or t30 = 30 minutes) in two different treatment periods in a cross-over manner. There will be 3 different cohorts with 2 treatment periods in each cohort.
  Interventions: Drug: Fast-acting insulin aspart; Device: iLet™

INTERVENTIONS:
Drug: Fast-acting insulin aspart — In each cohort, participants will receive fast-acting insulin aspart using the iLet™ in a cross-over manner for 14 days (7days per period). Dose modification will be handled autonomously by the iLet™ based on the CGM sensor readings and the user interaction with the iLet™ e.g. meal announcements.
Device: iLet™ — The bionic pancreas including pigtail adapters, used in insulin-only configuration

SUMMARY:
The iLet™ is a new insulin pump that is programmed to work with a Continuous Glucose Monitoring (CGM) device. This is to give participants insulin automatically. The CGM device is already available for sale. The iLet™ is not yet approved for use. Fast-acting insulin aspart is a type of insulin that doctors can already prescribe for use with insulin pens, but not for use in an insulin pump. This study is to test how safe fast acting insulin aspart is when used with different insulin delivery settings in the iLet™ in people with type 1 diabetes. Participants will get fast-acting insulin aspart as participants' insulin and use the iLet™ as participants' insulin pump with a CGM device. Participants' iLet™ will be set to 2 different insulin delivery settings for 7 days on each setting. The setting participants get first is decided by chance. The study will last for about 5 to 9 weeks. Participants will have 4 visits and 1 phone contact with the study or staff.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, age more than or equal to 18 years and less than or equal to 75 years at the time of signing informed consent
* Diagnosed with type 1 diabetes mellitus more than or equal to 1 year prior to the day of screening
* Treated with continuous subcutaneous insulin infusion more than or equal to 1 year prior to the day of screening
* Have a mean total daily dose of insulin more than or equal to 20 units
* Familiar with continuous glucose monitoring as judged by the investigator
* Has someone over 18 years of age who (i) lives with them, (ii) has access to where they sleep, (iii) is willing to be in the house when the subject is sleeping, and (iv) is willing to receive calls from the study staff and check the welfare of the study subject
* Body mass index (BMI) less than or equal to 35.0 kg/m^2 at screening
* Glycated haemoglobin (HbA1c) more than or equal to 6.5% (47 mmol/mol) and less than or equal to 9% (75 mmol/mol) at screening
* Able and willing to remain in a designated place for the specified duration of the 'in-patient' periods
* Lives within a 120-minute drive away from the central monitoring location (site)

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products
* Previous participation in this trial. Participation is defined as signed informed consent
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice)
* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days before screening
* Any disorder, except for conditions associated with diabetes mellitus, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Anticipated initiation or change in concomitant medications known to affect weight or glucose metabolism during the trial
* Impaired liver function, defined as Alanine Aminotransferase (ALT) more than or equal to 2.5 times or Bilirubin more than 1.5 times upper normal limit at screening
* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of eGFR less than 60 ml/min/1.73 m^2
* Any episodes of diabetic ketoacidosis within the past 90 days prior to the day of screening
* Known hypoglycaemic unawareness as indicated by the Investigator according to Clarke's questionnaire question 8
* Recurrent severe hypoglycaemic episodes within the last year as judged by the Investigator
* Any of the following: myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within the past 180 days prior to the day of screening
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Inadequately treated blood pressure defined as Grade 3 hypertension or higher (systolic more than or equal to 180 mmHg or diastolic more than or equal to 110 mmHg) at screening
* Unwilling or unable to avoid acetaminophen throughout the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results

REFERENCES:
- [Derived] Russell SJ, Balliro C, Ekelund M, El-Khatib F, Graungaard T, Greaux E, Hillard M, Jafri RZ, Rathor N, Selagamsetty R, Sherwood J, Damiano ER. Improvements in Glycemic Control Achieved by Altering the tmax Setting in the iLet(R) Bionic Pancreas When Using Fast-Acting Insulin Aspart: A Randomized Trial. Diabetes Ther. 2021 Jul;12(7):2019-2033. doi: 10.1007/s13300-021-01087-x. Epub 2021 Jun 19. PMID 34146238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at one site in the United States.
Groups:
- Cohort 1: t65 First, Then t50: iLet™ is a new insulin pump that is programmed to work with a Continuous Glucose Monitoring (CGM) device. Participants received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t50 = 50 minutes) for 7 days. The total treatment duration for each cohort was 14 days.
- Cohort 1: t50 First, Then t65: iLet™ is a new insulin pump that is programmed to work with a Continuous Glucose Monitoring (CGM) device. Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t50 = 50 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. The total treatment duration for each cohort was 14 days.
- Cohort 2: t65 First, Then t40; Cohort 3: t65 First, Then t30: iLet™ is a new insulin pump that is programmed to work with a Continuous Glucose Monitoring (CGM) device. Participants received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t40 = 40 minutes) for 7 days. The total treatment duration for each cohort was 14 days.
- Cohort 2: t40 First, Then t65: iLet™ is a new insulin pump that is programmed to work with a Continuous Glucose Monitoring (CGM) device. Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t40 = 40 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. The total treatment duration for each cohort was 14 days.
- Cohort 3: t30 First, Then t65: iLet™ is a new insulin pump that is programmed to work with a Continuous Glucose Monitoring (CGM) device. Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t30 = 30 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. The total treatment duration for each cohort was 14 days.
Period: First Treatment Period (7 Days)
Arm/Group | Cohort 1: t65 First, Then t50 | Cohort 1: t50 First, Then t65 | Cohort 2: t65 First, Then t40 | Cohort 2: t40 First, Then t65 | Cohort 3: t65 First, Then t30 | Cohort 3: t30 First, Then t65
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Second Treatment Period (7 Days)
Arm/Group | Cohort 1: t65 First, Then t50 | Cohort 1: t50 First, Then t65 | Cohort 2: t65 First, Then t40 | Cohort 2: t40 First, Then t65 | Cohort 3: t65 First, Then t30 | Cohort 3: t30 First, Then t65
Started | 4 | 4 | 4 | 4 | 4 | 3
Completed | 4 | 4 | 4 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Unclassified | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Participants were randomised in a 1:1 manner to one of two treatment sequences. First sequence: Participants received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t50 = 50 minutes) for 7 days. Second sequence: Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t50 = 50 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. The total treatment duration for the cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
- Cohort 2: Participants were randomised in a 1:1 manner to one of two treatment sequences. First sequence: Participants received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t40 = 40 minutes) for 7 days. Second sequence: Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t40 = 40 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. The total treatment duration for the cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
- Cohort 3: Participants were randomised in a 1:1 manner to one of two treatment sequences. First sequence: Participants received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t30 = 30 minutes) for 7 days. Second sequence: Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t30 = 30 minutes) for 7 days. After 7 days they received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) for 7 days. The total treatment duration for the cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (13.5) | 36.3 (14.8) | 47.1 (10.7) | 43.0 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 5 | 18
  Male | 2 | 1 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 8 | 8 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time in Low Interstitial Glucose (Defined as Below 54 mg/dL [3 mmol/L]) From Initiation of Treatment (Day 1) to End of Treatment (Day 7) (Percentage)
Description: Interstitial glucose: glucose measured in interstitial fluid. Time in low interstitial glucose (defined as below 54 mg/dL [3 mmol/L]) from initiation of treatment (day 1) to end of treatment (day 7). Time spent in low interstitial glucose is calculated as the percentage of available interstitial glucose values below the threshold.
Time Frame: Day 1 to day 7
Population: Full analysis set: included all randomised subjects receiving treatment.Number of participants analysed=participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- t50 Faster Aspart Cohort 1: Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t50 = 50 minutes) in cohort 1. The total treatment duration for each cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
- t65 Faster Aspart Cohort 1: Participants received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) in cohort 1. The total treatment duration for each cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
- t40 Faster Aspart Cohort 2: Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t40 = 40 minutes) in cohort 2. The total treatment duration for each cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
- t65 Faster Aspart Cohort 2: Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t65 = 65 minutes) in cohort 2. The total treatment duration for each cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
- t30 Faster Aspart Cohort 3: Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t30 = 30 minutes) in cohort 3. The total treatment duration for each cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
- t65 Faster Aspart Cohort 3: Participants received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) in cohort 3. The total treatment duration for each cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
Arm/Group | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 1 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 2 | t30 Faster Aspart Cohort 3 | t65 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7
Percentage | 0.98 (0.72) | 0.89 (1.16) | 0.69 (0.50) | 0.50 (0.79) | 0.61 (0.56) | 0.37 (0.41)

2. Primary Outcome: Time in Low Interstitial Glucose (Defined as Below 54 mg/dL [3 mmol/L]) From Initiation of Treatment (Day 1) to End of Treatment (Day 7) (Percentage) - Median
Description: as for outcome 1
Time Frame: Day 1 to day 7
Population: Full analysis set: included all randomised subjects receiving treatment. Number of participants analysed=participants with available data.
Measure: Median (Full Range); unit: Percentage
Arm/Group | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 1 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 2 | t30 Faster Aspart Cohort 3 | t65 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7
Percentage | 0.93 [0.2 to 2.2] | 0.42 [0.1 to 3.6] | 0.75 [0.0 to 1.4] | 0.20 [0.0 to 2.3] | 0.58 [0.0 to 1.4] | 0.29 [0.1 to 1.3]

3. Secondary Outcome: Number of Treatment Emergent Severe Hypoglycaemic Episodes
Description: Number of treatment emergent severe hypoglycaemic episodes from initiation of treatment (day 1) to end of treatment (day 7). Treatment emergent is defined as an episode that has onset in the period from initiation of treatment to end of treatment.
  Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective actions. Plasma glucose (PG) concentrations may not be available during an event, but neurological recovery following the return of PG to normal is considered sufficient evidence that the event was induced by a low PG concentration.
Time Frame: Day 1 to day 7
Population: Safety analysis set (SAS): included all subjects receiving treatment. Number of participants analysed=participants with available data.
Measure: Number; unit: Episodes
Groups:
- t50 Faster Aspart Cohort 2: Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t50 = 50 minutes) in cohort 2. The total treatment duration for each cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
Arm/Group | t50 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 1 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 2 | t30 Faster Aspart Cohort 3 | t65 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7
Episodes | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Self-manageable (Able to Self-treat) Treatment Emergent Hypoglycaemic Episodes That Require Oral Carbohydrate Intervention Per Day
Description: Mean number of self-manageable (able to self-treat) treatment emergent hypoglycaemic episodes that require oral carbohydrate intervention per day. Self-manageable (able to self-treat) hypoglycaemic episodes that require oral carbohydrate intervention per day is calculated as the sum of all hypoglycaemic episodes where the subject is able to self-treat and that require oral carbohydrate intervention divided by the actual duration of the treatment period in days. Treatment emergent is defined as an episode that has onset in the period from initiation of treatment to end of treatment.
Time Frame: Day 1 to day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Episodes
Groups:
- t40 Faster Aspart Cohort 1: Participants received fast-acting insulin aspart with the iLet™ having non-default tmax in the algorithm settings (t40 = 40 minutes) in cohort 2. The total treatment duration for each cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
Arm/Group | t50 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 1 | t40 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 2 | t30 Faster Aspart Cohort 3 | t65 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7
Episodes | 1.01 (0.44) | 0.87 (0.49) | 1.06 (0.57) | 0.68 (0.43) | 0.86 (0.55) | 0.51 (0.36)

5. Secondary Outcome: Number of Treatment Emergent Overall Hypoglycaemic Episodes Classified According to the American Diabetes Association (ADA) Definition
Description: ADA classification of hypoglycaemia:
  1. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective actions.
  2. Asymptomatic hypoglycaemia: An episode not accompanied by typical symptoms of hypoglycaemia, but with a measured PG concentration ≤3.9 mmol/L (70 mg/dL).
  3. Documented symptomatic hypoglycaemia: An episode during which typical symptoms of hypoglycaemia are accompanied by a measured PG concentration ≤ 3.9 mmol/L (70 mg/dL).
  4. Pseudo-hypoglycaemia: An episode during which the person with diabetes reports any of the typical symptoms of hypoglycaemia with a measured PG concentration > 3.9 mmol/L (70 mg/dL) but approaching that level.
  5. Probable symptomatic hypoglycaemia: An episode during which symptoms of hypoglycaemia are not accompanied by a PG determination but that was presumably caused by a PG concentration ≤ 3.9 mmol/L (70 mg/dL).
Time Frame: Day 1 to day 7
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | t65 Faster Aspart Cohort 1 | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 2 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 3 | t30 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8
Episodes
  Severe hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 0
  Documented symptomatic hypoglycaemia | 36 | 38 | 24 | 42 | 17 | 25
  Asymptomatic hypoglycaemia | 9 | 15 | 8 | 6 | 4 | 9
  Probable symptomatic hypoglycaemia | 4 | 2 | 3 | 3 | 1 | 5
  Pseudo-hypoglycaemia | 3 | 8 | 3 | 6 | 3 | 6

6. Secondary Outcome: Number of Treatment Emergent Overall Hypoglycaemic Episodes Classified According to the Novo Nordisk Classification
Description: Overall hypoglycaemia count according to Novo Nordisk classification. Novo Nordisk classification of hypoglycaemia:
  1. Severe hypoglycaemia according to the ADA classification.
  2. Symptomatic BG confirmed hypoglycaemia: An episode that is BG confirmed by PG value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
  3. Asymptomatic BG confirmed hypoglycaemia: An episode that is BG confirmed by PG value <3.1 mmol/L (56 mg/dL) without symptoms consistent with hypoglycaemia.
  4. BG confirmed hypoglycaemia: The union of 2. and 3.
  5. Severe or BG confirmed symptomatic hypoglycaemia: The union of 1. and 2.
  6. Severe or BG confirmed hypoglycaemia: The union of 1., 2. and 3.
Time Frame: Day 1 to day 7
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | t65 Faster Aspart Cohort 1 | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 2 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 3 | t30 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8
Episodes
  Severe hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 0
  Symptomatic BG confirmed hypoglycaemia | 13 | 12 | 4 | 13 | 6 | 10
  Asymptomatic BG confirmed hypoglycaemia | 3 | 3 | 3 | 1 | 1 | 2
  BG confirmed hypoglycaemia | 16 | 15 | 7 | 14 | 7 | 12
  Severe or BG confirmed symptomatic hypoglycaemia | 13 | 12 | 4 | 13 | 6 | 10
  Severe or BG confirmed hypoglycaemia | 16 | 15 | 7 | 14 | 7 | 12

7. Secondary Outcome: Number of Treatment Emergent Daytime Hypoglycaemic Episodes Classified According to the American Diabetes Association (ADA) Definition
Description: as for outcome 5
Time Frame: Day 1 to day 7 (in both the treatment periods)
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | t65 Faster Aspart Cohort 1 | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 2 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 3 | t30 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8
Episodes
  Severe hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 0
  Documented symptomatic hypoglycaemia | 30 | 31 | 21 | 35 | 14 | 22
  Asymptomatic hypoglycaemia | 5 | 11 | 5 | 4 | 4 | 7
  Probable symptomatic hypoglycaemia | 3 | 2 | 3 | 2 | 0 | 4
  Pseudo-hypoglycaemia | 2 | 5 | 3 | 6 | 2 | 6

8. Secondary Outcome: Number of Treatment Emergent Daytime Hypoglycaemic Episodes Classified According to the Novo Nordisk Classification
Description: Number of daytime hypoglycaemic episodes according to Novo Nordisk classification. Novo Nordisk classification of hypoglycaemia:
  1. Severe hypoglycaemia according to the ADA classification.
  2. Symptomatic BG confirmed hypoglycaemia: An episode that is BG confirmed by PG value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
  3. Asymptomatic BG confirmed hypoglycaemia: An episode that is BG confirmed by PG value <3.1 mmol/L (56 mg/dL) without symptoms consistent with hypoglycaemia.
  4. BG confirmed hypoglycaemia: The union of 2. and 3.
  5. Severe or BG confirmed symptomatic hypoglycaemia: The union of 1. and 2.
  6. Severe or BG confirmed hypoglycaemia: The union of 1., 2. and 3.
Time Frame: Day 1 to day 7
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | t65 Faster Aspart Cohort 1 | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 2 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 3 | t30 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8
Episodes
  Severe hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 0
  Symptomatic BG confirmed hypoglycaemia | 12 | 9 | 3 | 9 | 3 | 9
  Asymptomatic BG confirmed hypoglycaemia | 2 | 1 | 2 | 0 | 1 | 2
  BG confirmed hypoglycaemia | 14 | 10 | 5 | 9 | 4 | 11
  Severe or BG confirmed symptomatic hypoglycaemia | 12 | 9 | 3 | 9 | 3 | 9
  Severe or BG confirmed hypoglycaemia | 14 | 10 | 5 | 9 | 4 | 11

9. Secondary Outcome: Number of Treatment Emergent Nocturnal Hypoglycaemic Episodes Classified According to the American Diabetes Association (ADA) Definition
Description: as for outcome 5
Time Frame: Day 1 to day 7
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | t65 Faster Aspart Cohort 1 | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 2 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 3 | t30 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8
Episodes
  Severe hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 0
  Documented symptomatic hypoglycaemia | 6 | 7 | 3 | 7 | 3 | 3
  Asymptomatic hypoglycaemia | 4 | 4 | 3 | 2 | 0 | 2
  Probable symptomatic hypoglycaemia | 1 | 0 | 0 | 1 | 1 | 1
  Pseudo-hypoglycaemia | 1 | 3 | 0 | 0 | 1 | 0

10. Secondary Outcome: Number of Treatment Emergent Nocturnal Hypoglycaemic Episodes Classified According to the Novo Nordisk Classification
Description: Number of nocturnal (from time 00:01-05:59 both inclusive) hypoglycaemic episodes according to Novo Nordisk classification. Novo Nordisk classification of hypoglycaemia:
  1. Severe hypoglycaemia according to the ADA classification.
  2. Symptomatic BG confirmed hypoglycaemia: An episode that is BG confirmed by PG value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
  3. Asymptomatic BG confirmed hypoglycaemia: An episode that is BG confirmed by PG value <3.1 mmol/L (56 mg/dL) without symptoms consistent with hypoglycaemia.
  4. BG confirmed hypoglycaemia: The union of 2. and 3.
  5. Severe or BG confirmed symptomatic hypoglycaemia: The union of 1. and 2.
  6. Severe or BG confirmed hypoglycaemia: The union of 1., 2. and 3.
Time Frame: Day 1 to day 7 (in both the treatment periods)
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | t65 Faster Aspart Cohort 1 | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 2 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 3 | t30 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8
Episodes
  Severe hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 0
  Symptomatic BG confirmed hypoglycaemia | 1 | 3 | 1 | 4 | 3 | 1
  Asymptomatic BG confirmed hypoglycaemia | 1 | 2 | 1 | 1 | 0 | 0
  BG confirmed hypoglycaemia | 2 | 5 | 2 | 5 | 3 | 1
  Severe or BG confirmed symptomatic hypoglycaemia | 1 | 3 | 1 | 4 | 3 | 1
  Severe or BG confirmed hypoglycaemia | 2 | 5 | 2 | 5 | 3 | 1

11. Secondary Outcome: Time in Interstitial Glucose Range Was Defined as 70-180 mg/dL (3.9-10 mmol/L) From Initiation of Treatment (Day 1) to End of Treatment (Day 7) (Percentages)
Description: Time in interstitial glucose range defined as 70-180 mg/dL (3.9-10 mmol/L) from initiation of treatment (day 1) to end of treatment (day 7). Time spent in interstitial glucose range is calculated as the percentage of available interstitial glucose values above or equal to the low threshold and below or equal to the high threshold.
Time Frame: Day 1 to day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 1 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 2 | t30 Faster Aspart Cohort 3 | t65 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7
Percentage | 70.87 (9.35) | 66.79 (10.39) | 73.93 (6.14) | 70.44 (8.49) | 78.32 (6.96) | 73.82 (11.79)

12. Secondary Outcome: Mean Interstitial-glucose Level
Description: Mean interstitial glucose level is calculated as the average of the available interstitial glucose values.
Time Frame: Day 1 to day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 1 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 2 | t30 Faster Aspart Cohort 3 | t65 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7
mg/dL | 150.3 (7.8) | 157.7 (11.0) | 150.1 (8.5) | 157.6 (11.5) | 144.1 (7.1) | 152.5 (11.4)

13. Secondary Outcome: Number of Treatment Emergent Adverse Events
Description: Number of treatment emergent adverse events from initiation of treatment (day 1) to end of treatment (day 7). Treatment emergent is defined as an event that has onset in the period from initiation of treatment to end of treatment.
Time Frame: Day 1 to day 7
Population: as for outcome 3
Measure: Number; unit: Events
Arm/Group | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 1 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 2 | t30 Faster Aspart Cohort 3 | t65 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7
Events | 2 | 2 | 2 | 0 | 0 | 1

14. Secondary Outcome: Number of Treatment Emergent Infusion Site Reactions
Description: Number of treatment-emergent infusion site reactions from initiation of treatment (day 1) to end of treatment (day 7). Treatment emergent is defined as an event that has onset in the period from initiation of treatment to end of treatment.
Time Frame: Day 1 to day 7
Population: as for outcome 3
Measure: Number; unit: Infusion site reaction
Arm/Group | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 1 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 2 | t30 Faster Aspart Cohort 3 | t65 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7
Infusion site reaction | 0 | 0 | 0 | 0 | 0 | 1

15. Secondary Outcome: Total Insulin Dose Per Day
Description: Total insulin dose (U/kg) per day from initiation of treatment (day 1) to end of treatment (day 7). Total daily insulin dose is calculated as the sum of all insulin doses delivered by the iLet™ divided by the actual duration of the treatment period in days.
Time Frame: Day 1 to day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/Kg/day
Arm/Group | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 1 | t40 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 2 | t30 Faster Aspart Cohort 3 | t65 Faster Aspart Cohort 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7
U/Kg/day | 0.60 (0.12) | 0.63 (0.12) | 0.65 (0.13) | 0.67 (0.16) | 0.63 (0.12) | 0.64 (0.18)

ADVERSE EVENTS:
Time Frame: From the first trial-related activity (screening, day -14) after obtaining informed consent and until the follow up visit (treatment days 7 in both periiods+7 days follow-up)
Description: All adverse events listed are treatment emergent. Treatment emergent is defined as an event that has onset in the period from initiation of treatment to end of treatment.
Groups:
- t65 Faster Aspart Cohort 2: Participants received fast-acting insulin aspart with the iLet™ having default tmax in the algorithm settings (t65 = 65 minutes) in cohort 2. The total treatment duration for each cohort was 14 days with each cross-over period of the 2 tmax settings being 7 days.
Arm/Group | t50 Faster Aspart Cohort 1 | t65 Faster Aspart Cohort 1 | t40 Faster Aspart Cohort 2 | t65 Faster Aspart Cohort 2 | t30 Faster Aspart Cohort 3 | t65 Faster Aspart Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 2/8 | 1/8 | 1/8 | 0/8 | 0/8 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | t50 Faster Aspart Cohort 1 (N=8) | t65 Faster Aspart Cohort 1 (N=8) | t40 Faster Aspart Cohort 2 (N=8) | t65 Faster Aspart Cohort 2 (N=8) | t30 Faster Aspart Cohort 3 (N=8) | t65 Faster Aspart Cohort 3 (N=7)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT03816761/Prot_SAP_000.pdf